CLINICAL TRIAL: NCT03607110
Title: Comparison of Ketamine-propofol Sedation Protocols With Fentanyl-propofol Administered by Endoscopist or Anesthesiologist at Colonoscopy
Brief Title: Comparison of Efficacy of Anesthesia Administered by Endoscopist or Anesthesiologist on Colonoscopy
Status: Completed | Type: Observational
Sponsor: Selda KAYAALTI (Other Government)
Responsible Party: Sponsor-Investigator, Selda KAYAALTI, Anesthesia and Reanimation Specialist, Develi Devlet Hastanesi
Organization: Develi Devlet Hastanesi (Other Government)
Other Study IDs: 2018/94
Record Dates: First submitted 2018-07-13; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Colonoscopy; Ketamine; Fentanyl
MeSH Terms: interventions — Ketamine; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- ketamine: ketamine used
  Interventions: Drug: Ketamine; Device: patient control analgesia
- fentanyl: fentanyl used
  Interventions: Drug: fentanyl; Device: patient control analgesia

INTERVENTIONS:
Drug: Ketamine — sedation drugs
  Groups: ketamine
Drug: fentanyl — sedation drugs
  Groups: fentanyl
Device: patient control analgesia — patient control analgesia

SUMMARY:
In sedation applications performed by an endoscopist or anesthetist during colonoscopy, it was investigated whether there were differences in pain levels evaluated by VAS (Visuel analog scale), patient satisfaction, duration of procedure and side effects

DETAILED DESCRIPTION:
Gastrointestinal endoscopes are an invasive and unpleasant procedure that is increasingly being performed worldwide (1). Colonoscopy; is one of the endoscopic procedures that can be used to diagnose and treat large intestine and cause pain and excessive discomfort in the patient (2). For this reason, intravenous (iv) sedative agents are used in endoscopy centers where endoscopy will be performed. However, side effects such as hypoxia and hypotension, which are usually dose-dependent, caused by these sedative agents, play an important role among risk factors associated with colonoscopy (3). For this reason, the use of propofol as an anesthetic is prohibited in some countries, which is a commonly used agent for sedation. However, the presence of an anesthetist during each endoscopy procedure is difficult because there are not enough anesthetists. This application is also more costly. For this reason, studies have been carried out during the gastrointestinal endoscopy when sedation is delivered by someone other than the anesthetist (4). For this purpose, several studies comparing patient-controlled sedation or sedation applied by an endoscopist to sedation performed by anesthesiologist were performed (4, 5). Investigators aimed to investigate whether there is any difference between the two groups in terms of pain levels assessed by VAS (Visuel analog scale) and patient satisfaction by comparing sedation protocols applied by endoscopist or anesthesist during colonoscopy in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accept the method and will undergo elective colonoscopy
* ASA I-II group
* Patients with the ability to perform VAS scoring

Exclusion Criteria:

* Patients who do not accept the method
* ASA III-IV-V group of patients with uncontrolled chronic disease (such as uncontrolled hypertension, uncontrolled diabetes mellitus)
* Patients with severe respiratory failure and cardiovascular disease
* Patients with liver and kidney failure
* Patients with long-term analgesic, opioid, sedative use history - Patients who are known to be hypersensitive to study medications, eggs,
* Those who are of pregnancy or pregnancy and those who are in breastfeeding period
* Those with antipsychotic or antidepressant medication usage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colonoscopy patients with ASA I-II group
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
pain level - VAS SCALE | during the operation
  Pain level assessed by VAS
patient satisfaction - Patient satisfaction Scale | during the operation
  patient satisfaction assessed by with satisfaction score of 4 points-scale (1 very good, 2 good, 3 not bad, 4 bad)

SECONDARY OUTCOMES:
operation time | during the operation
  duration of operation time will be asssessed as min.
side effects questionnaire | during the operation
  Cardio pulmonary side effects (Hypotension, Bradycardia, Desaturation) and other side effects (Nausea and Vomiting, Headache)

CONTACTS AND LOCATIONS:
Locations (1):
- Develi Hatice Muammer Kocatürk Devlet Hastanesi, Develi, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Ferreira AO, Cravo M. Sedation in gastrointestinal endoscopy: Where are we at in 2014? World J Gastrointest Endosc. 2015 Feb 16;7(2):102-9. doi: 10.4253/wjge.v7.i2.102. PMID 25685266
- [Background] Dal H., S. İzdeş, E. Kesimci, et al. Kolonoskopide sedasyon için propofolün aralıklı bolus veya hedef kontrollü infüzyon yöntemiyle uygulanmasının karşılaştırılması, Türk Anest Rean Der Dergisi, 2011; 39(3): 134-142
- [Background] Lee DW, Chan AC, Sze TS, Ko CW, Poon CM, Chan KC, Sin KS, Chung SC. Patient-controlled sedation versus intravenous sedation for colonoscopy in elderly patients: a prospective randomized controlled trial. Gastrointest Endosc. 2002 Nov;56(5):629-32. doi: 10.1067/mge.2002.128919. PMID 12397267
- [Background] Poincloux L, Laquiere A, Bazin JE, Monzy F, Artigues F, Bonny C, Abergel A, Dapoigny M, Bommelaer G. A randomized controlled trial of endoscopist vs. anaesthetist-administered sedation for colonoscopy. Dig Liver Dis. 2011 Jul;43(7):553-8. doi: 10.1016/j.dld.2011.02.007. Epub 2011 Mar 29. PMID 21450542
- [Background] Crepeau T, Poincloux L, Bonny C, Lighetto S, Jaffeux P, Artigue F, Walleckx P, Bazin JE, Dapoigny M, Bommelaer G. Significance of patient-controlled sedation during colonoscopy. Results from a prospective randomized controlled study. Gastroenterol Clin Biol. 2005 Nov;29(11):1090-6. doi: 10.1016/s0399-8320(05)82172-4. PMID 16505753